CLINICAL TRIAL: NCT01305135
Title: A Phase I-II Study of the Efficacy and Safety of Idarubicin Combined to Azacitidine in Int-2 or High Risk Myelodysplastic Syndromes
Brief Title: Idarubicin Combined to Azacitidine in Int-2 or High Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-AZA-IDA-09
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: High Grade Myelodysplastic Syndrome Lesions
Keywords: myelodysplastic syndrome, azacitidine, idarubicin
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azacitidine 75mg/m²/d + idarubicin 5mg/m²/d (Experimental): phase I : palier 1 have 10 patients and palier 2 have to 10 patients.
  palier 1: Ida 5mg/m²/d (D8) + AZACITIDINE 75mg/m²/d (D1-D7)
  Interventions: Drug: azacitidine and idarubicin
- Azacitidine 75mg/m²/d + idarubicin 10mg/m²/d (Experimental): palier 2: Ida 10mg/m²/d (D8)+ Azacitidine 75mg/m²/d (D1-D7)
  Interventions: Drug: azacitidine and idarubicin

INTERVENTIONS:
Drug: azacitidine and idarubicin — azacitidine:100mg, 75mg/m²/d, during 7days every 28 days (D1-D7). Idarubicin: 5mg/ml, 5mg/m²/d (palier1) or 10mg/m²/d (palier2), D8

SUMMARY:
Patients will receive escalating doses of ldarubicin combined to Azacitidine given at the FDA/EMEA approved Schedule and dosing.

For the Phase I study :

Determine the safety and tolerance of escalating doses of Idarubicin combined to Azacitidine in patients with INT-2 or higher risk MDS.

For the phase II study:

Primary: Evaluate rate and duration of response (according to IWG 2006 criteria and IWG 2000 criteria) to the combination of Idarubicin and Azacitidine in patients with INT-2 or higher risk MDS

DETAILED DESCRIPTION:
Patients will receive ldarubicin combined to Azacitidine.

* The first 10 patients will receive Idarubicin 5 mg/m2/d on day 8 of each cycle of Azacitidine 75 mg/m2/d CI during 7 days (First Cohort ).
* Progression or not to the next cohort of 10 patients : Idarubicin 10 mgm2/d on day 8 of each cycle of Azacitidine 75 mg/m2/d CI during 7 days (Second cohort of 10 patients), will be decided after completion of the first cohort, after review of hematological toxicity by an independent safety review committee (SRC).
* The next 21 patients will be treated either according to the first or second cohort schedule of Idarubicin, after review of hematological toxicity and efficacy by an independent safety review committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MDS, or CMML with WBC < 13,000/mm3 that meets IPSS criteria for intermediate-2 or high-risk disease,
* IPSS score ≥1.5
* Myocardial function do not contraindicate the use of idarubicin
* Age ≥ 18 years
* Performance Status ≤2 according to ECOG.
* Serum creatinine < 1.5 x ULN and normal levels of electrolytes (serum sodium 136-145 mmol/l, Potassium 3,5-4,5 mmol/l, alkaline Reserve 23-29 mmol/l, , Calcium 2,15-2,5 mmol/l, Phosphore 0,87-1,45 mmol/l) Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) < 1.5 x upper limit of normal (ULN)
* Serum total bilirubin < 1.5 x ULN.
* Must be able to adhere to the study visit schedule and other protocol requirements
* Signed informed consent.

Female subjects of childbearing potential must:

• Accept effective contraception without interruption throughout the duration of study and up to three months after the end of treatment.

Male subjects must

* Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy and up to three months after the final treatment if their partner is of childbearing potential and has no contraception.
* Agree to learn the procedures for preservation of sperm

Exclusion Criteria:

* Uncontrolled infection
* Prior therapy with anthracycline for MDS.
* Eligible for an allogeneic stem cell transplantation.
* Prior therapy with demethylating agents within the last 3 months
* Prior therapy with Hematopoietic growth factor (ESA or G-CSF) agents or cytotoxic agents (oral chemotherapy, low doses AraC) within the last 30 days.
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast)
* Pregnant or lactating females
* Known HIV-1 positivity
* Contra-indication to Anthracyclines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12-30 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2016-05-09 (Actual)

PRIMARY OUTCOMES:
To determined tolerance and dose limiting toxicities to idarubicin and azacitidine association. | After 12 weeks treatment

SECONDARY OUTCOMES:
to determined overall response rate and response duration | After six months

CONTACTS AND LOCATIONS:
Overall Officials: Lionel ADES, PHD,MD, Principal Investigator — GFM: Groupe Francophone des Myélodysplasies
Locations (32):
- France (31):
  - CHU de Haut-Lévèque, Pessac, Bordeaux - Pessac
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - Hôpital de la cote basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHRU de Caen - Hôpital Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - CHU Dijon Hôpital d'enfants, Dijon
  - CHU Albert Michallon, Grenoble
  - CH Le Mans, Le Mans
  - CHU de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli-Calmette, Marseille
  - CHU Brabois, Nancy
  - CHU Hotel dieu, Nantes
  - CHU NICE, Hôpital l'Archet, Nice
  - Hôpital saint louis - Hématologie Clinique, Paris
  - Hôpital Saint Louis - Hématologie Séniors, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital cochin, Paris
  - Centre hospitalier Joffre, Perpignan
  - CH de Périgueux, Périgueux
  - CHU de Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital Hautepierre, Strasbourg
  - Hôpital PURPAN - Hématologie Clinique, Toulouse
  - Hôpital Purpan - Médecine Interne, Toulouse
  - Hôpital Bretonneau, Tours
  - CH de Valence, Valence
  - Institut Gustave Roussy, Villejuif
- Hôpital Aziza Othmana, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No